CLINICAL TRIAL: NCT00063440
Title: Epidemiology of Carotid IMT Progression in MESA - Ancillary Study
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1214; 5R01HL069003-05 (NIH)
Record Dates: First submitted 2003-06-26; First posted 2003-06-30 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Carotid Artery Diseases; Coronary Arteriosclerosis
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Carotid Artery Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To determine the factors associated with progression of sub-clinical atherosclerosis and to evaluate the associations between the progression of sub-clinical atherosclerosis and the development of clinically manifest atherosclerosis.

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease remains the leading cause of death in the United States and one of the leading causes of morbidity. New technology recently has allowed the non-invasive investigation of the extent of atherosclerosis in different vascular beds. Unfortunately, the clinical implications and significance of this new technology have not yet been fully examined nor has the interrelationship between these various measurements of clinical and sub-clinical atherosclerosis. The study is ancillary to the Multi-Ethnic Study of Atherosclerosis (MESA), an NHLBI-supported epidemiological study of atherosclerosis in several ethnic groups.

DESIGN NARRATIVE:

A longitudinal assessment of the carotid intima media thickness (IMT) will be added to the scheduled follow-up visits in MESA subjects in order to study the relationship between carotid IMT and a measure of calcium burden in the coronary vessels. In addition, studies will be conducted on how these two non-invasive markers of atherosclerosis relate to cardiovascular disease risk factors and clinical events.The study will utilize the MESA cohort involving 6500 subjects who will have baseline and four follow-up examinations. coronary artery calcification (CAC) and IMT are being obtained at baseline, with CAC determinations also scheduled at follow-up. IMT determinations will be added in conjunction with the CAC studies in the second and third exams and detailed analyses will be carried out on these two measures of atherosclerotic burden that may reflect different biologic processes.

ELIGIBILITY:
Members of MESA study

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the Multi-Ethnic Study of Atherosclerosis, a cross-sectional NIH population cohort originating from 6 regions in the United States
Sampling Method: Non-Probability Sample
Enrollment: 5610 (Actual)
Dates: Start 2003-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Common carotid artery intima-media thickness | randomly selected at 2 years or 4 years in 1/2 of the cohort

SECONDARY OUTCOMES:
Common carotid artery diameter | randomly selected at 2 or 4 years for each 1/2 of the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Polak, MD, MPH, Principal Investigator — Tufts Medical Center

REFERENCES:
- [Derived] Polak JF, Herrington D, O'Leary DH. Associations of edge-detected and manual-traced common carotid artery intima-media thickness with incident peripheral artery disease: The Multi-Ethnic Study of Atherosclerosis. Vasc Med. 2019 Aug;24(4):306-312. doi: 10.1177/1358863X19835925. Epub 2019 Apr 26. PMID 31023166
- [Derived] Polak JF, O'Leary DH. Edge-detected common carotid artery intima-media thickness and incident coronary heart disease in the multi-ethnic study of atherosclerosis. J Am Heart Assoc. 2015 Jun 15;4(6):e001492. doi: 10.1161/JAHA.114.001492. PMID 26077584
- [Derived] Polak JF, Sacco RL, Post WS, Vaidya D, Arnan MK, O'Leary DH. Incident stroke is associated with common carotid artery diameter and not common carotid artery intima-media thickness. Stroke. 2014 May;45(5):1442-6. doi: 10.1161/STROKEAHA.114.004850. Epub 2014 Mar 18. PMID 24643408
- [Derived] Polak JF, Johnson C, Harrington A, Wong Q, O'Leary DH, Burke G, Yanez ND. Changes in carotid intima-media thickness during the cardiac cycle: the multi-ethnic study of atherosclerosis. J Am Heart Assoc. 2012 Aug;1(4):e001420. doi: 10.1161/JAHA.112.001420. Epub 2012 Aug 24. PMID 23130162
- [Derived] Polak JF, Wong Q, Johnson WC, Bluemke DA, Harrington A, O'Leary DH, Yanez ND. Associations of cardiovascular risk factors, carotid intima-media thickness and left ventricular mass with inter-adventitial diameters of the common carotid artery: the Multi-Ethnic Study of Atherosclerosis (MESA). Atherosclerosis. 2011 Oct;218(2):344-9. doi: 10.1016/j.atherosclerosis.2011.05.033. Epub 2011 Jun 14. PMID 21726862